CLINICAL TRIAL: NCT03639597
Title: Clinical Investigation of the VytronUS Ablation System for Treatment of Paroxysmal Atrial Fibrillation - The VALUE Study
Brief Title: Clinical Investigation of the VytronUS Ablation System for Treatment of Paroxysmal Atrial Fibrillation
Acronym: VALUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VytronUS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 980-06114-00
Record Dates: First submitted 2018-07-17; First posted 2018-08-21 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: ablation; ultrasound; automation; catheter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study device (Experimental): VytronUS Ablation System
  Interventions: Device: VytronUS Ablation System

INTERVENTIONS:
Device: VytronUS Ablation System

SUMMARY:
The study is a single center, open-label, single arm, prospective pre-market study designed to assess the safety and efficacy of the VytronUS Ablation System (VAS) for the treatment of atrial fibrillation in patients with drug refractory, recurrent, symptomatic, paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Subjects with documented symptomatic, recurrent, PAF refractory to at least one beta blocker, calcium channel blocker or Class I or Class III anti-arrhythmic drug, who meet all inclusion/exclusion criteria and are deemed appropriate candidates for catheter ablation will undergo PV ablation with the VAS. Pre-procedural CT scan or MRI will be obtained to assess LA and PV anatomy and size. PV ablation will be performed utilizing the VAS (see procedure description below). Acute post-ablation confirmation of PV electrical isolation will be evaluated via standard mapping techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. History of symptomatic recurrent paroxysmal atrial fibrillation (PAF) in the prior year, defined by:

   a.Episodes of AF i.≥2 recurrent AF episodes of more than 30 seconds' duration that self-terminate and lasting no more than 7 continuous days or ii.Episodes of AF ≤ 48 hours duration terminated with electrical or pharmacologic cardioversion count as a paroxysmal atrial fibrillation episode b.At least one episode of paroxysmal atrial fibrillation (PAF) documented on 12-lead ECG, event monitor, or telemetry monitor in the prior year
3. Paroxysmal atrial fibrillation refractory to at least one Beta Blocker, Calcium Channel Blocker, or Class I or Class III anti-arrhythmic drug (AAD).
4. Subject is indicated for a pulmonary vein ablation according to society guidelines or investigational site practice.
5. Subject is able and willing to give informed consent.
6. Willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full duration of the study.

Exclusion Criteria:

1. Non-paroxysmal AF (e.g. persistent, long-standing persistent, or permanent AF)
2. AF secondary to electrolyte imbalance, thyroid disease or reversible or non-cardiac cause.
3. Prior LA ablation or surgery
4. Women known to be pregnant or breastfeeding or of childbearing potential unless on satisfactory contraceptive routine
5. NYHA Class III or IV congestive heart disease
6. LVEF <40% measured by acceptable cardiac testing (eg. TTE, TEE)
7. Anteroposterior LA diameter >5.5cm or <3.0cm by TTE
8. Presence of intracardiac thrombus (including a known history of thrombus) within 30 days prior to the index ablation procedure
9. Presence of pulmonary vein stent(s)
10. Presence of pre-existing pulmonary narrowing or pulmonary vein stenosis
11. Presence of a cardiac valve prosthesis
12. Bleeding diathesis or contraindication to anticoagulation therapy
13. Blood clotting abnormalities (genetic)
14. MI, PCI, invasive cardiac procedure or surgery within 90 days prior to the index ablation procedure
15. Previous CVA, TIA, or PE within 3 months prior to the index procedure
16. Structural heart defect that, in the investigator's opinion, prevents catheter access or increases risk of ablation procedure
17. Pacemaker, ICD, or CRT implantation within 6 months prior to the index ablation procedure
18. Active systemic infection
19. Subject contraindicated for both MRI and CT
20. Life expectancy less than 360 days in physician's opinion
21. Participation in a drug or device study
22. Exclusion as per local laws -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy - Acute success and chronic freedom from AF, AFL and AT lasting longer than 30 seconds, freedom from new class I or II AAD | 12 months
  Acute (or technical) procedural success defined as PVI documented by confirmed entrance block. Chronic success defined by freedom from symptomatic AF, AT and AFL lasting longer than 30 seconds, freedom from new class I or II AAD and no repeat ablation through 12 months of follow-up.
Primary Safety - incidence of acute AEs occurring within 7 days of procedure and chronic adverse events | 12 months
  Acute major AEs occurring within 7 days of procedure and chronic AEs defined as symptomatic PV stenosis >70% or symptomatic atrio-esophageal fistula diagnosed within 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Na Homolce, Prague, Czechia

REFERENCES:
- [Derived] Turagam MK, Petru J, Neuzil P, Kakita K, Kralovec S, Harari D, Phillips P, Piazza D, Whang W, Dukkipati SR, Reddy VY. Automated Noncontact Ultrasound Imaging and Ablation System for the Treatment of Atrial Fibrillation: Outcomes of the First-in-Human VALUE Trial. Circ Arrhythm Electrophysiol. 2020 Mar;13(3):e007917. doi: 10.1161/CIRCEP.119.007917. Epub 2020 Feb 12. PMID 32078362